CLINICAL TRIAL: NCT03112434
Title: Use of Elastography to Quantify Change in Upper Extremity Muscle Spasticity Following Botox Injection in Children With Spastic Cerebral Palsy
Brief Title: Muscle Elastography in Spastic Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Radiological Society of North America (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-628
Record Dates: First submitted 2017-04-03; First posted 2017-04-13 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Unilateral Spastic Cerebral Palsy
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Botulinum toxin type A — Botox injection in upper extremity for spasticity in pediatric CP patients

SUMMARY:
To date, clinical tests are unable to differentiate between the cause of muscle stiffness, although a manual instrumented spasticity assessment for the lower limb that utilizes surface electromyogram has recently been proposed. This study intends to use shear wave elastography to assess individual muscle stiffness parameters and the individual response to botulinum toxin injection in the elbow and wrist flexors. Collection of baseline spasticity parameters could then be used to predict the effect of botulinum toxin type A and ultimately serve as a basis for development of a treatment model for muscle spasticity in patients with spastic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral spastic cerebral palsy with presence of dynamic muscle spasticity in the elbow and/or wrist flexors, who will be able to provide consent.
* Consent may be obtained from a parent or legal guardian, as applicable.

Exclusion Criteria:

* Prior surgical procedure in the affected upper extremity
* Unrelated orthopedic injury to the affected upper extremity
* Current oral or intrathecal antispasticity therapy
* Prior Botulinum toxin type A injection in preceding 6 months

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with unilateral spastic CP with presence of dynamic muscle spasticity in the elbow and/or wrist flexors, who will be able to provide consent. Consent may be obtained from a parent or legal guardian, as applicable.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Muscle Elasticity | From immediate pre-injection to 1 month post-injection.
  Change in muscle elasticity (in kilopascal )
Muscle Elasticity | From immediate pre-injection to 1 month post-injection.
  Change in muscle elasticity (in m/s)

SECONDARY OUTCOMES:
Functional measures | immediately pre- and immediately post-injection, and at 1 month, 3 months and 6 months post-injection.
  Functional measures (MAS)
Functional measures | immediately pre- and immediately post-injection, and at 1 month, 3 months and 6 months post-injection.
  Functional measures (PROM)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No